CLINICAL TRIAL: NCT01692444
Title: Role of Fibrocytes in the Bronchial Remodelling of Chronic Obstructive Pulmonary Disease
Acronym: FIBROCHIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2011/34
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Fibrosis; Fibroblast; Lung attenuation; Pletysmography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung tissue form surgery such as lobectomy or pneumonectomy,whole blood sample for fibrocytes analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- COPD: 15 patients with COPD from 1 to 4 according to the GOLD 2011
- Non smoker Control: 15 patients without COPD and no smoking history
- Smoker Control: 15 patients without COPD but a smoking history

SUMMARY:
Airway remodelling is an abnormal tissue repair following bronchial inflammation, which contributes to none reversible pathological features, such as bronchial and peri-bronchial fibrosis. It also influences the prognosis of Chronic Obstructive Pulmonary Disease (COPD) and its mechanisms remain largely unknown. The role of fibrocytes has been demonstrated in the pathophysiology of asthma, lung fibrosis or pulmonary hypertension. However, the recruitment of blood fibrocytes and their involvement in COPD airway remodelling remain unknown.

The main objective of the study is to analyse the distribution and quantify the number of the peri-bronchial and blood circulating fibrocytes in patients with different stages of COPD compared to control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 40 yr
* Patient needed a thoracic surgery such as lobectomy for cancer or lung transplantation or lung reduction volume surgery.
* COPD group: diagnostic of COPD and differentiation of the stage from 1 to 4 according to the GOLD guidelines.
* Control group: subjects with normal lung function testing and no chronic symptoms (cough or expectoration). Subjects will be separated in 2 groups according to smoking history (Never smokers, smokers (former or current) and paired to patients according to age and sex.
* with a written informed consent

Exclusion Criteria:

* Subject without any social security or health insurance
* Asthma, lung fibrosis or idiopathic pulmonary hypertension
* Chronic viral infections (hepatitis, HIV)
* Pregnant woman or breastfeeding
* Subject included for cancer surgery with a Pn0 diagnosis not confirmed after the intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Controls and COPD patients will be recruited during surgical visit or hospitalization in thoracic surgery department before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Increased number of peri-bronchial and blood circulating fibrocytes gradually in each stages of COPD and compared to control subjects. | Lung tissues and blood samples will be collected at inclusion visit during surgery (Day 0)

SECONDARY OUTCOMES:
Characterization of fibrocytes: expression of chemokines receptors, Toll Like Receptors, HLA class II | Lung tissues and blood samples will be collected at inclusion visit during surgery (Day 0)
Correlation between lung attenuation and the number of fibrocytes | Assessed one year after inclusion visit (i.e. surgery date =Day 0)
Correlation between plethysmography and the number of fibrocytes. | Assessed one year after inclusion visit (i.e. surgery date = Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas MOORE, MD-PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- University hospital of Bordeaux, Hôpital du Haut Lévêque, Pessac, France

REFERENCES:
- [Derived] Eyraud E, Maurat E, Sac-Epee JM, Henrot P, Zysman M, Esteves P, Trian T, Dupuy JW, Leipold A, Saliba AE, Begueret H, Girodet PO, Thumerel M, Hustache-Castaing R, Marthan R, Levet F, Vallois P, Contin-Bordes C, Berger P, Dupin I. Short-range interactions between fibrocytes and CD8+ T cells in COPD bronchial inflammatory response. Elife. 2023 Jul 26;12:RP85875. doi: 10.7554/eLife.85875. PMID 37494277
- [Derived] Henrot P, Beaufils F, Thumerel M, Eyraud E, Boudoussier A, Begueret H, Maurat E, Girodet PO, Marthan R, Berger P, Dupin I, Zysman M. Circulating fibrocytes as a new tool to predict lung cancer progression after surgery? Eur Respir J. 2021 Dec 9;58(6):2101221. doi: 10.1183/13993003.01221-2021. Print 2021 Dec. No abstract available. PMID 34561289